CLINICAL TRIAL: NCT04383080
Title: The Effect and Safety of Low-level Laser Therapy in Acute Decompensated Heart Failure Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NYMUH IRB No.2019b007
Record Dates: First submitted 2020-04-30; First posted 2020-05-11 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Acupuncture
Keywords: Low-level Laser; Acupuncture therapy; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Acupuncture Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-level laser therapy (Experimental): Low-level laser irradiation on specific acupuncture points
  Interventions: Device: Low-level laser therapy
- Acupuncture therapy (Active Comparator): Dry needle inserting specific acupuncture points
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — acupuncture at specific acupuncture points
  Arms: Acupuncture therapy
Device: Low-level laser therapy — low level laser emission on specific acupuncture points
  Arms: Low-level laser therapy

SUMMARY:
The advantages of laser acupuncture are a non-invasive, painless, low risk of infection and high safety. Laser acupuncture as a treatment tool has the following advantages1.Painless, 2. Non-invasive treatment, the subject is highly accepted, the risk of infection and needle stick is low, 3. Very few side effects such as fainting, bleeding, 4. The therapeutic dose is easy to operate, and the instrument output frequency, power and time can be controlled. Through the clinical physiological function test plus the verification and analysis of the quantitative test values, it will be more able to define the new role of laser acupuncture treatment in patients with heart failure from the perspective of Chinese medicine.

DETAILED DESCRIPTION:
From the perspective of ancient books, the discussion of heart failure in the etiology and pathogenesis of traditional Chinese medicine was first seen in the "Shu Wen". It is clearly pointed out that "heart qi" is the basic pathogenesis of heart failure. The "qi" and "blood" of Chinese medicine are closely related. The blood line is driven by the gas, the blood is bloody, and the qi deficiency is unable to push the blood to blood. If the qi deficiency, it would lead to blood stasis; There were studies have indicated that traditional acupuncture treatment can increase exercise tolerance and adjust autonomic nerve activity in patients with chronic heart failure, and can reduce their readmission rate and mortality rate in patients with acute heart failure. Studies using laser acupuncture to treat patients with heart failure have also found that they can increase the subject's six-minute walking distance.

ELIGIBILITY:
Inclusion Criteria:

* Age over 20 years of age, with written informed consent.
* NYHA:stage II-III.
* All patients had LVEF <40% caused by dilated or ischemic cardiomyopathy.
* Acute HF patient presenting with dyspnea related to cardiogenic pulmonary edema.
* All patients had sinus rhythm, were stable and compensated with individually optimized standard heart failure medication as well as oral anticoagulants for at least 3 months before (including prophylactic defibrillator placement).
* Systolic blood pressure > 95 mmHg at admission.
* B-type natriuretic peptide (BNP) > 150 pg/mL or NT-pro BNP > 600 pg/mL.

Exclusion Criteria:

* Age under 20.
* Major cardiovascular events and treatments occurred four weeks before hospitalization.
* Major cardiovascular surgery or treatment will be performed in the next 6 months.
* Pregnant or expected to pregnancy within a year.
* Require a heart transplant in 6 months.
* Uncontrolled atrial or ventricular dysrhythmias.
* Uncompensated congestive heart failure.
* Heart failure due to congenital heart disease or obstructive myocardial disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
N- terminal pro-brain natriuretic peptide, NT-proBNP | At the 12th week and 24th week
  The change of NT-pro BNP from the date of admission to the end of trial

SECONDARY OUTCOMES:
High sensitivity C-Reactive Protein, hs-CRP Hs-CRP | At the 12th week and 24th week
  The change of NT-pro BNP from the date of admission to the end of trial

OTHER OUTCOMES:
Questionnaires_Instrumental activities of daily living | At the 4th, 12t, 20th and 24th week
  (IADL);Scoring from 0 to 4 and higher scores mean better outcome.
Questionnaires_EuroQol- 5 Dimension | At the 4th, 12t, 20th and 24th week
  (EQ-5D);Scoring from 1 to 3 and higher scores mean better outcome.
Questionnaires_The Minnesota LIVING WITH HEART FAILURE® Questionnaire | At the 4th, 12t, 20th and 24th week
  (MLHFQ);Scoring from 0 to 5 and higher scores mean better outcome.
Questionnaires_Patient Health Questionnaire-9 | At the 4th, 12t, 20th and 24th week
  (PHQ-9);Scoring from 0 to 3 and higher scores mean worse outcome.
Questionnaires_Constitution in Chinese Medicine Questionnaire | At the 4th, 12th, 20th and 24th week
  (CCMQ);Scoring from 1 to 5 and higher scores correspond to specific body constitution.
6 minutes walking test | At the 4th, 12t, 20th and 24th week
  (6 minutes walking distance, meters)
Left ventricular ejection fraction | At the 24th week
  (Ejection fraction, %)
Heart rate variability_SDNN | At the 12th and 24th week
  (Standard deviation of all normal to normal intervals, ms)
Heart rate variability_SDANN index | At the 12th and 24th week
  (Standard deviation of average normal to normal intervals index, ms)
Heart rate variability_ASDNN | At the 12th and 24th week
  (Average standard deviation of all 5-min R-R intervals, ms)
Heart rate variability_rMSSD | At the 12th and 24th week
  (The square root of the mean of the sum of the squares of differences between adjacent NN intervals, ms)
Heart rate variability_LF | At the 12th and 24th week
  (Low frequency power, normalized unit/ n.u. and ms2)
Heart rate variability_HF | At the 12th and 24th week
  (High frequency power, normalized unit/ n.u. and ms2)
Heart rate variability_LF/HF | At the 12th and 24th week
  (LF/HF Ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Shih Meng Chu, Bachelor, Principal Investigator — National Yang Ming Chiao Tung University Hospital
Locations (1):
- National Yang Ming University Hospital, Yilan, Taiwan